CLINICAL TRIAL: NCT00948922
Title: Evaluation of Melphalan+Bortezomib as a Conditioning Regimen for Autologous and Allogeneic Stem Cell Transplants in Multiple Myeloma After Cytoreductive Therapy
Brief Title: Melphalan+Bortezomib as a Conditioning Regimen for Autologous and Allogeneic Stem Cell Transplants in Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: H. Lee Moffitt Cancer Center and Research Institute (Other)
Collaborators: Millennium Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MCC-15697; XO5271 (Other Grant/Funding Number: Millennium)
Record Dates: First submitted 2009-07-28; First posted 2009-07-29 (Estimated); Results first posted 2018-10-12 (Actual); Last update posted 2019-09-18 (Actual); Status verified 2019-06

CONDITIONS: Multiple Myeloma
Keywords: multiple myeloma; myeloma; myeloma proteins; autologous; allogeneic; G-CSR; granulocyte colony-stimulating factor; stem cell transplant; stem cell; stem cell mobilization
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — Bortezomib; Melphalan; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- A: Allogeneic Stem Cell Transplant (Other): Allogeneic Stem Cell Transplant: Fludarabine+Melphalan+Bortezomib followed by Allogeneic Rescue.
  Interventions: Drug: Bortezomib; Drug: Melphalan; Drug: Fludarabine; Procedure: Allogeneic Stem Cell Transplant
- B: Autologous Stem Cell Transplant (Other): Autologous Stem Cell Transplant: Melphalan+Bortezomib followed by Autologous Rescue.
  Interventions: Drug: Bortezomib; Drug: Melphalan; Procedure: Autologous Stem Cell Transplant
- BE: Group B Expansion (Other): Group B Expansion on Bortezomib Maintenance: Autologous Only.
  Interventions: Drug: Bortezomib; Drug: Melphalan; Procedure: Autologous Stem Cell Transplant

INTERVENTIONS:
Drug: Bortezomib — AUTOLOGOUS ARM: Day -3 bortezomib (1.3 mg/m^2) as an intravenous push over 3 to 5 seconds (follows Melphalan infusion). ALLOGENEIC ARM: Day -3 bortezomib (1.3 mg/m^2) as an intravenous push over 3 to 5 seconds (follows fludarabine and melphalan infusion).
  Other Names: Velcade
Drug: Melphalan — AUTOLOGOUS ARM: Day -4 and Day -3 Melphalan 100 mg/m^2/day IV over 30 minutes. ALLOGENEIC ARM: Day -4, Day -3 Melphalan 70 mg/m^2/day IV over 30 minutes.
  Other Names: Alkeran(R)
Procedure: Autologous Stem Cell Transplant — Autologous Stem Cell Transplant: Autologous Peripheral Blood Stem Cell Rescue. Stem cell mobilization with granulocyte colony-stimulating factor (GCSF) at a dose of 10 μg/kg/day as per institutional standards. CD34+ peripheral blood stem cells will be collected following the administration of G-CSF as per institutional standards. Day 0 Infusion of autologous stem cells.
  Arms: B: Autologous Stem Cell Transplant; BE: Group B Expansion
Drug: Fludarabine — Days -6,-5,-4,-3 Fludarabine 30 mg/m^2/day IV
  Other Names: Fludara(R)
  Arms: A: Allogeneic Stem Cell Transplant
Procedure: Allogeneic Stem Cell Transplant — Allogeneic Stem Cell Transplant: Allogeneic Peripheral Blood Stem Cell Rescue. Day 0 Infusion of allogeneic peripheral blood stem cells. For the allogeneic matched-related donors peripheral blood stem cells will be harvested with GCSF mobilization and infused fresh to the recipients. Allogeneic donor stem cells may also be cryopreserved if they cannot be infused fresh.
  Arms: A: Allogeneic Stem Cell Transplant

SUMMARY:
The purpose of this study is to evaluate the effectiveness of Bortezomib when added to standard chemotherapy medicine(s) for treatment of Multiple Myeloma.

DETAILED DESCRIPTION:
The primary objectives of this study are:

* To determine the 2 year-progression free survival in multiple myeloma with an allogeneic transplant using a conditioning regimen of melphalan + fludarabine + Bortezomib in patients < 60 years of age and available HLA-matched donor and compare it with the 2 year-progression-free-survival after an autologous stem cell transplant with melphalan+Bortezomib conditioning in patients < 60 years.
* To determine the 2 year-progression free survival in multiple myeloma with an autologous stem cell transplant using a conditioning regimen of melphalan + Bortezomib. for patients > 60 years of age and patients < 60 years of age who decline allogeneic stem cell transplant.

The secondary objectives of this study are:

* To determine the overall survival in multiple myeloma with autologous or allogeneic stem cell transplants using the above conditioning regimens
* To determine the response rates in multiple myeloma using the above regimens.
* To determine minimal residual disease status using allele specific oligonucleotides (ASO-PCR) by PCR and flow-cytometry for multiple myeloma cells.
* To correlate minimal residual disease status with 2 year progression free survival and overall survival.
* To determine the incidence of acute and chronic graft-versus-host disease (GVHD) in multiple myeloma with allogeneic stem cell transplant using the above conditioning regimen.
* To examine quality of life in patients treated with allogeneic and autologous stem cell transplants using the above conditioning regimen.

ELIGIBILITY:
Inclusion Criteria:

Multiple Myeloma Criteria(International Uniform Response Criteria for Multiple Myeloma)

* Patients with responsive disease after any line of induction therapy
* A complete response
* A very good partial response
* A partial response
* Patients greater than or equal to 18 years of age are eligible. There is upper age limit of 60 years for allogeneic transplants.
* Patients must have a histologically confirmed diagnosis.
* All patients should have a life expectancy of at least 12 weeks.
* Patients must have undergone a complete psychosocial evaluation and have been considered capable of compliance.
* Meet the following criteria for allogeneic hematopoietic cell transplant:
* Must have an identified donor match defined as: HLA-A, HLA-B, HLA- C, DRB1 8/8 allele matched sibling, family member, or unrelated donor. [7/8 would go on separate mismatched trials] and be < 60 years of age.
* Calculated hematopoietic cell transplantation-specific comorbidity index (HCT-CI) <3

Exclusion Criteria:

* Patients who do not achieve at least a partial response (PR) by the criteria mentioned above with induction therapy.
* Patient has a platelet count of <30 x 10^9/L within 14 days before enrollment.
* Patient has >/= Grade 2 peripheral neuropathy within 30 days before enrollment.
* Patient has an absolute neutrophil count of <1.0 x 10^9/L within 30 days before enrollment.
* Myocardial infarction within 6 months prior to enrollment or has New York Hospital Association (NYHA) Class III or IV heart failure, uncontrolled angina, severe uncontrolled ventricular arrhythmias, or electrocardiographic evidence of acute ischemia or active conduction system abnormalities. Prior to study entry, any ECG abnormality at screening has to be documented by the investigator as not medically relevant in order for the subject to be considered eligible. Left ventricular ejection fraction (LVEF) by multiple gated acquisition (MUGA) scan < 40%.
* Patient has hypersensitivity to bortezomib, boron or mannitol.
* Female subject is pregnant or breast-feeding. Confirmation that the subject is not pregnant must be established by a negative serum beta-human chorionic gonadotropin (beta-hCG) pregnancy test result obtained during screening. Pregnancy testing is not required for post-menopausal or surgically sterilized women.
* Patient has received other investigational drugs with 30 days before enrollment
* Serious medical or psychiatric illness likely to interfere with participation in this clinical study.
* Patients with a diffusing capacity of lung for carbon monoxide (DLCO) less than 50% (adjusted) of normal or with symptomatic obstructive or restrictive lung disease are ineligible.
* Patients with a total bilirubin greater than 2.0 mg/dL excluding Gilbert's syndrome and serum glutamate oxaloacetate transaminase (SGOT) or serum glutamate pyruvate transaminase (SGPT) greater than two and a half times normal (unless due to primary malignancy), or a history of severe hepatic dysfunction are ineligible.
* Calculated creatinine clearance </= 30 ml/min within 30 days before enrollment
* Patients with active infections are ineligible.
* Patients who are HIV positive are ineligible.
* Patients with active leptomeningeal involvement are ineligible. Patients with a history of previous cerebrospinal fluid (CSF) tumor involvement without symptoms or signs are eligible provided the CSF is now free of disease on lumbar puncture, and MRI of the brain shows no tumor involvement. Patients with severe symptomatic central nervous system (CNS) disease of any etiology are ineligible.
* Patients with uncontrolled insulin-dependent diabetes mellitus defined as a random glucose level of > 400 in the 30 days prior to initiation of study therapy; or uncompensated major thyroid or adrenal dysfunction are ineligible.
* Patients with an Eastern Cooperative Oncology Group (ECOG) performance status of >/= 2(Karnofsky < 50%) are ineligible.
* Patients with an ECOG performance status of 2 to 3(Karnofsky 30-50%), secondary to bone pain, may be enrolled.
* Patients with an ECOG performance status of 2 to 3(Karnofsky 30-50%), secondary to a potentially reversible disease-related problem, may be enrolled.
* Patients with any previous malignancy other than non-melanoma skin cancer are ineligible, unless the patient is without evidence of disease >/= 5 years after the treatment for the cancer was completed.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 124 (Actual)
Dates: Start 2009-06-18 (Actual); Primary Completion 2017-04-20 (Actual); Study Completion 2019-05-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Alsina, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute; Jose Ochoa-Bayona, MD, Principal Investigator — H. Lee Moffitt Cancer Center and Research Institute
Locations (1):
- H. Lee Moffitt Cancer Center, Tampa, Florida, United States

REFERENCES:
- See also: H. Lee Moffitt Cancer Center & Research Institute website — http://www.moffitt.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at Moffitt Cancer Center August 2009 through April 2015.
Groups:
- A: Allogeneic Stem Cell Transplant: Allogeneic Stem Cell Transplant: Fludarabine+Melphalan+Bortezomib followed by Allogeneic Rescue.
  Bortezomib: AUTOLOGOUS ARM: Day -3 bortezomib (1.3 mg/m^2) as an intravenous push over 3 to 5 seconds (follows Melphalan infusion). ALLOGENEIC ARM: Day -3 bortezomib (1.3 mg/m^2) as an intravenous push over 3 to 5 seconds (follows fludarabine and melphalan infusion).
  Melphalan: AUTOLOGOUS ARM: Day -4 and Day -3 Melphalan 100 mg/m^2/day IV over 30 minutes. ALLOGENEIC ARM: Day -4, Day -3 Melphalan 70 mg/m^2/day IV over 30 minutes.
  Fludarabine: Days -6,-5,-4,-3 Fludarabine 30 mg/m^2/day IV
  Allogeneic Stem Cell Transplant: Allogeneic Peripheral Blood Stem Cell Rescue. Day 0 Infusion of allogeneic peripheral blood stem cells. For the allogeneic matched-related donors peripheral blood stem cells will be harvested with granulocyte colony-stimulating factor (GCSF) mobilization and infused fresh to recipients. Allogeneic donor stem cells may be cryopreserved if they cannot be infused
- B: Autologous Stem Cell Transplant: Autologous Stem Cell Transplant: Melphalan+Bortezomib followed by Autologous Rescue.
  Bortezomib: AUTOLOGOUS ARM: Day -3 bortezomib (1.3 mg/m^2) as an intravenous push over 3 to 5 seconds (follows Melphalan infusion). ALLOGENEIC ARM: Day -3 bortezomib (1.3 mg/m^2) as an intravenous push over 3 to 5 seconds (follows fludarabine and melphalan infusion).
  Melphalan: AUTOLOGOUS ARM: Day -4 and Day -3 Melphalan 100 mg/m^2/day IV over 30 minutes. ALLOGENEIC ARM: Day -4, Day -3 Melphalan 70 mg/m^2/day IV over 30 minutes.
  Autologous Stem Cell Transplant: Autologous Stem Cell Transplant: Autologous Peripheral Blood Stem Cell Rescue. Stem cell mobilization with granulocyte colony-stimulating factor (G-CSF) at a dose of 10 μg/kg/day as per institutional standards. CD34+ peripheral blood stem cells will be collected following the administration of G-CSF as per institutional standards. Day 0 Infusion of autologous stem cells.
- BE: Group B Expansion: Group B Expansion on Bortezomib Maintenance: Autologous Only.
  Bortezomib: AUTOLOGOUS ARM: Day -3 bortezomib (1.3 mg/m^2) as an intravenous push over 3 to 5 seconds (follows Melphalan infusion). ALLOGENEIC ARM: Day -3 bortezomib (1.3 mg/m^2) as an intravenous push over 3 to 5 seconds (follows fludarabine and melphalan infusion).
  Melphalan: AUTOLOGOUS ARM: Day -4 and Day -3 Melphalan 100 mg/m^2/day IV over 30 minutes. ALLOGENEIC ARM: Day -4, Day -3 Melphalan 70 mg/m^2/day IV over 30 minutes.
  Autologous Stem Cell Transplant: Autologous Stem Cell Transplant: Autologous Peripheral Blood Stem Cell Rescue. Stem cell mobilization with granulocyte colony-stimulating factor (G-CSF) at a dose of 10 μg/kg/day as per institutional standards. CD34+ peripheral blood stem cells will be collected following the administration of G-CSF as per institutional standards. Day 0 Infusion of autologous stem cells.
Period: Overall Study
Arm/Group | A: Allogeneic Stem Cell Transplant | B: Autologous Stem Cell Transplant | BE: Group B Expansion
Started | 34 | 51 | 39
Completed | 26 | 37 | 38
Not Completed | 8 | 14 | 1
Not completed — Did not start study treatment | 2 | 5 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 1
Not completed — Death | 3 | 0 | 0
Not completed — Disease progression | 0 | 1 | 0
Not completed — Insurance issues | 1 | 0 | 0
Not completed — Transplant eligibility issues | 2 | 3 | 0
Not completed — Not evaluable at time of analysis | 0 | 3 | 0

BASELINE CHARACTERISTICS:
Population: Baseline: All participants enrolled on study. Adverse Events: All participants who received study treatment. Outcome Measures: All participants evaluable at time of analysis.
Groups:
- Total: Total of all reporting groups
Arm/Group | A: Allogeneic Stem Cell Transplant | B: Autologous Stem Cell Transplant | BE: Group B Expansion | Total
Number analyzed (Participants) | 34 | 51 | 39 | 124
Age, Continuous [Mean (Full Range); unit: years] | 53.5 [32 to 76] | 62 [31 to 79] | 62 [39 to 78] | 60 [31 to 79]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 20 | 19 | 62
  Male | 11 | 31 | 20 | 62
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 8 | 9 | 19
  Not Hispanic or Latino | 32 | 43 | 29 | 104
  Unknown or Not Reported | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 1 | 1
  Asian | 1 | 1 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 1 | 7 | 3 | 11
  White | 32 | 38 | 32 | 102
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 5 | 3 | 8
Region of Enrollment [Number; unit: participants]
  United States | 34 | 51 | 39 | 124

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS: Number of participants, per treatment arm with progression free survival at time of analysis. Survival time will be measured from the date of transplant to the date of progression, death or the last follow-up, whichever comes first. Progressive Disease (PD): Increase of ≥ 25% from lowest response value in any one or more of the following: Serum M-component and/or; Urine M-component and/or; Only in patients without measurable serum and urine M-protein levels; the difference between involved and uninvolved FLC levels. The absolute increase must be > 10 mg/dL; Bone marrow plasma cell percentage; absolute percentage ≥ 10%; Definite development of new bone lesions or soft tissue plasmacytomas or definite increase in the size of existing bone lesions or soft tissue plasmacytomas; Development of hypercalcemia that can be attributed solely to the plasma cell proliferative disorder.
Time Frame: End of 2 year, post transplant follow-up
Population: All participants evaluable at time of analysis
Measure: Count of Participants; unit: Participants
Arm/Group | A: Allogeneic Stem Cell Transplant | B: Autologous Stem Cell Transplant | BE: Group B Expansion
Number analyzed (Participants) | 26 | 37 | 38
Participants | 17 | 25 | 19

2. Secondary Outcome: Overall Survival (OS) Rate
Description: Overall survival in participants with multiple myeloma treated with Bortezomib (Velcade®) containing conditioning regimen and autologous as well as allogeneic transplantation.
Time Frame: End of 2 year, post transplant follow-up
Measure: Number (95% Confidence Interval); unit: percentage
Arm/Group | A: Allogeneic Stem Cell Transplant | B: Autologous Stem Cell Transplant | BE: Group B Expansion
Number analyzed (Participants) | 26 | 37 | 38
percentage | 79.2 [57.0 to 90.8] | 89.2 [73.7 to 95.8] | 97.3 [82.3 to 99.6]

3. Secondary Outcome: Molecular Complete Response (CR) Rates in Patients With Multiple Myeloma
Description: Complete Response according to International Myeloma Working Group uniform response criteria. CR: Negative immunofixation on the serum and urine and disappearance of any soft tissue plasmacytomas and < 5% plasma cells in bone marrow.
Time Frame: End of 2 year, post transplant follow-up
Population: Patients were in very good partial response at the time on enrollment without sufficient plasma cells in bone marrow to be able to perform assay for molecular response.
Arm/Group | A: Allogeneic Stem Cell Transplant | B: Autologous Stem Cell Transplant | BE: Group B Expansion
Number analyzed (Participants) | 0 | 0 | 0

4. Other Pre Specified Outcome: Percentage of Participants With Acute or Chronic Graft-versus-host Disease (GVHD) Following Transplant
Description: Percentage of participants with Acute or Chronic GVHD following transplant
Time Frame: End of 2 year, post transplant follow-up
Population: Allogenic Stem Cell Transplant patients only. Autologous patients do not suffer from GVHD.
Measure: Number; unit: percentage of participants
Groups:
- A: Allogenic Stem Cell Transplant: Allogenic Stem Cell Transplant: Fludarabine + Melphalan + Bortezomib followed by Allogenic Rescue
Arm/Group | A: Allogenic Stem Cell Transplant
Number analyzed (Participants) | 26
percentage of participants | 34

ADVERSE EVENTS:
Time Frame: 7 years, 8 months
Description: All Serious Adverse Events are reported, regardless of causality. For this study that includes patients undergoing hematopoietic cell transplantation (HCT), review and consideration was given for reporting of Other Adverse Events that are designated in the protocol as commonly observed after HCT. Patients are monitored for Serious Adverse Events and Other Adverse events beginning at on treatment date. Patients who did not receive treatment: not included in at risk numbers.
Arm/Group | A: Allogeneic Stem Cell Transplant | B: Autologous Stem Cell Transplant | BE: Group B Expansion
All-Cause Mortality (participants affected / at risk) | 3/32 | 1/42 | 0/39
Serious Adverse Events (participants affected / at risk) | 13/32 | 18/42 | 10/39
Other Adverse Events (participants affected / at risk) | 0/32 | 1/42 | 0/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Allogeneic Stem Cell Transplant (N=32) | B: Autologous Stem Cell Transplant (N=42) | BE: Group B Expansion (N=39)
Allergic reaction (Immune system disorders) | 0 (0) | 1 (1) | 0 (0)
Blood/Bone Marrow - Other (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
Haptoglobin (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Hemolysis (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)
Neutrophil count decreased (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 2 (2)
Supraventricular and nodal arrhythmia - Atrial fibrillation (Cardiac disorders) | 0 (0) | 3 (3) | 0 (0)
Cardiac General - Other (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
Cardiopulmonary arrest, cause unknown (non-fatal) (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1)
Hypotension (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
Fatigue (General disorders) | 0 (0) | 1 (1) | 0 (0)
Fever (in the absence of neutropenia) (General disorders) | 3 (3) | 0 (0) | 0 (0)
Death not associated with CTCAE term (General disorders) | 3 (3) | 1 (1) | 0 (0)
Dehydration (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Dysphagia (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Esophagitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Gastrointestinal - Other (Gastrointestinal disorders) | 1 (1) | 1 (1) | 0 (0)
Mucositis/stomatitis (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | 2 (2)
Typhlitis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1) | 1 (2)
Hemorrhage/Bleeding - Other, knee effusion (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Colitis, infectious (Infections and infestations) | 0 (0) | 1 (1) | 1 (1)
Febrile neutropenia (Infections and infestations) | 1 (1) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Brain (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Lung (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Paranasal (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Salivary gland (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection with normal ANC or Grade 1 or 2 neutrophils - Skin (Infections and infestations) | 0 (0) | 0 (0) | 1 (1)
Infection with unknown ANC - Appendix (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection with unknown ANC - Gallbladder (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Infection with unknown ANC - Salivary gland (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
Infection with unknown ANC - Skin (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
Opportunistic infection associated with >= Grade 2 Lymphopenia (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
ALT, SGPT - Increase (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
AST, SGOT - Increase (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Alkaline phosphatase (Metabolism and nutrition disorders) | 1 (1) | 1 (1) | 0 (0)
Calcium, serum-high (hypercalcemia) (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0)
Arthritis (non-septic) (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0)
Ataxia (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)
Extrapyramidal/involuntary movement/restlessness (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
Mental status (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
Pain - Back (Musculoskeletal and connective tissue disorders) | 1 (1) | 1 (1) | 0 (0)
Bronchospasm, wheezing (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 1 (1) | 0 (0)
Edema, larynx (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | 0 (0)
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary/Upper Respiratory - Other, Pneumonia (Respiratory, thoracic and mediastinal disorders) | 1 (2) | 0 (0) | 0 (0)
Pulmonary/Upper Respiratory - Other, Pulmonary edema (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
Pulmonary/Upper Respiratory - Other, Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1)
Renal failure (Renal and urinary disorders) | 2 (2) | 1 (1) | 2 (2)
Renal/Genitourinary - Other, Renal insufficiency (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
Renal/Genitourinary - Other, Hematuria (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1)
Secondary malignancy - possibly related to cancer treatment (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0)
Thrombosis/embolism (vascular access-related) (Vascular disorders) | 1 (1) | 1 (1) | 0 (0)
Thrombosis/thrombus/embolism (Vascular disorders) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A: Allogeneic Stem Cell Transplant (N=32) | B: Autologous Stem Cell Transplant (N=42) | BE: Group B Expansion (N=39)
Lymphopenia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | 0 (0)

LIMITATIONS AND CAVEATS:
SAEs not recorded for participants off study, though they were followed for survival.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-06-09): https://cdn.clinicaltrials.gov/large-docs/22/NCT00948922/Prot_SAP_000.pdf